CLINICAL TRIAL: NCT05776628
Title: Evaluation of the Performance and Safety of Plenum® Tissue Ortho for the Prevention of Epidural Fibrosis and Post-laminectomy Syndrome After Microdiscectomy, for the Treatment of Disc Herniation
Brief Title: Evaluation of Plenum® Tissue Ortho to Prevent Epidural Fibrosis and Post-laminectomy Syndrome.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: M3 Health (Industry)
Collaborators: Irmandade da Santa Casa de Misericordia de Sao Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Regenerative membrane; U1111-1302-0033 (Registry Identifier: UTN)
Record Dates: First submitted 2023-02-27; First posted 2023-03-20 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-11

CONDITIONS: Herniated Disk Lumbar

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polydioxanone membrane (Active Comparator): After flavectomy and manipulation of the spinal nerve and dura mater to resect the herniated intervertebral disk, the membrane will be placed on top of the dura mater.
  Interventions: Device: Plenum® Tissue ortho membrane (polydioxanone membrane)
- Control (No Intervention): The microdiscectomy procedure will be performed routinely, without the addition of any device over the dura mater.

INTERVENTIONS:
Device: Plenum® Tissue ortho membrane (polydioxanone membrane) — Membrane addition after flavectomy and spinal nerve and dura mater manipulation.
  Arms: Polydioxanone membrane

SUMMARY:
The goal of this clinical trial is to compare if adding a polydioxanone membrane prevents epidural fibrosis and, consequently, the rate of occurrence of the post-laminectomy syndrome in participants undergoing microdiscectomy for treatment of disc herniation.

DETAILED DESCRIPTION:
Participants will be submitted to microdiscectomy with the addition of a polydioxanone membrane over the dura mater in the test group and without in the control group.

The groups will be compared regarding improving patients' quality of life, evaluation of epidural fibrosis, and device safety.

ELIGIBILITY:
Inclusion Criteria:

* Pain radiating to one of the legs confirmed with an MRI scan;
* Patients who have already undergone conservative treatment (treatment with medication and physiotherapy) for at least 6 weeks, but have not shown improvement;
* Non-pregnant women or women of childbearing age who use contraceptive methods;
* Having signed the free and informed consent form (TCLE).

Exclusion Criteria:

* Patients with concomitant pathologies (eg infection or tumor and segmental instability or vertebral fractures);
* Cauda equina syndrome;
* Strength deficit characterized by strength equal to or less than III/V;
* Previous surgery of the lumbar spine;
* Patientes who have wound healing disorders;
* Patients with contraindications for evaluating MRI with the use of contrast;
* More than 1 herniated disk.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Patient's quality of life | Change from the baseline, to immediate potostoperative period (14 days) and to late postoperative period (6 months).
  Assessed by the Oswestry Questionnaire for lumbar evaluation (The low back pain disability Oswestry questionnaire).

SECONDARY OUTCOMES:
Epidural fibrosis | 6 months postoperatively.
  Evaluation of epidural fibrosis using Magnetic Resonance Imaging (IMR) will grade the scar from 0 to 4 for 5 contiguous axial slices centered around the intervertebral disc. The scar will be graded as none (0) (no scar on the dural surface), mild (1) (scar on less than 25% of the surface), mild-moderate (2) (scar on 25-50 % of the surface), (3) moderate-extensive (scarring on 50-75% of the surface), or extensive (4) (scarring on more than 75% of the surface).
Patient's quality of life | Before the procedure, in the immediate postoperative period (14 days) and in the late postoperative period (6 months).
  SF-36 Questionnaire
Low back and leg pain | Before the procedure, in the immediate postoperative period (14 days) and in the late postoperative period (6 months).
  Pain change will be measured by a Visual Analogue Scale (VAS)
Intervention safety | Through study completion, an average of 6 months
  Adverse events occurrence

CONTACTS AND LOCATIONS:
Overall Officials: Sybele Saska Specian, PhD, Study Director — M3 Health
Locations (1):
- M3 Health, Jundiaí, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No